CLINICAL TRIAL: NCT06225765
Title: A Prospective Trial Comparing Transoral Endoscopic Thyroidectomy Vestibular Approach (TOETVA) and Conventional Open Thyroidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tseung Kwan O Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, YEUNG WING CHI ZENON, Consultant, Department of Otorhinolaryngology, Head and Neck Surgery, Tseung Kwan O Hospital, Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC/KE-23-0006/FR-4
Record Dates: First submitted 2024-01-09; First posted 2024-01-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Benign Thyroid Nodule; Suspicious Malignant Thyroid Nodule
Keywords: Thyroid nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Prospective case control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transoral endoscopic thyroidectomy vestibular approach (TOETVA) (Experimental): Test group receiving surgery under transoral endoscopic thyroidectomy vestibular approach (TOETVA)
  Interventions: Procedure: Transoral endoscopic thyroidectomy vestibular approach (TOETVA)
- Traditional open surgery (Active Comparator): Control group receiving traditional open thyroidectomy
  Interventions: Procedure: Traditional Open Thyroidectomy

INTERVENTIONS:
Procedure: Transoral endoscopic thyroidectomy vestibular approach (TOETVA) — Remote access thyroid surgery
  Arms: Transoral endoscopic thyroidectomy vestibular approach (TOETVA)
Procedure: Traditional Open Thyroidectomy — Open thyroidectomy via trans-cervical approach
  Arms: Traditional open surgery

SUMMARY:
To determine if transoral endoscopic thyroidectomy vestibular approach (TOETVA) is a safe and effective procedure compared to traditional open thyroidectomy. Surgical outcomes, patients' satisfaction, voice and swallowing outcomes will be assessed.

DETAILED DESCRIPTION:
This is a prospective case control study involving a total 40 patients, with 20 stratified into the test group receiving surgery under transoral endoscopic thyroidectomy vestibular approach (TOETVA) and 20 patients to the control group under traditional open approach. Subjects will be assigned to either group without randomization. Patients satisfactory score, voice and swallowing quality of life outcomes will be assessed using Voice Handicap Index (VHI) and MD Anderson Dysphagia Inventory (MDADI) outcomes. Surgical outcomes, for instance, lower lip numbness, skin injury, operative time, blood loss, vocal cord paralysis, temporary and permanent hypoparathyroidism will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Benign thyroid nodule less than 4cm
* Suspicious malignant thyroid nodule less than 2cm, suitable for transoral endoscopic surgery

Exclusion Criteria:

* Patients under 18 years old
* Contraindication to general anaesthesia
* Vulnerable population (e.g. Cognitive impairment, pregnant)
* Previous anterior neck surgery
* Previous radiotherapy at the head and neck region
* Malignant thyroid nodule > 2cm
* Presence of another malignancy, lateral neck, or distant metastasis
* Retrosternal goitre
* Cervical spine disease precluding extension of the neck
* Obesity with BMI > 35kg/m2
* Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
* Untreated active infection
* Non-correctable coagulopathy
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient's satisfactory score | Post-operative day 1
  Visual analogue scale 0-10
Patient's satisfactory score | Post-operative 2 weeks
  Visual analogue scale 0-10
Patient's satisfactory score | Post-operative 6 months
  Visual analogue scale 0-10
Post-operative pain | Post-operative day 1
  Visual analogue scale 0-10
Post-operative pain | Post-operative 2 weeks
  Visual analogue scale 0-10
Post-operative pain | Post-operative 6 months
  Visual analogue scale 0-10
Voice quality of life | Post-operative day 1
  Voice Handicap Index - 30 assessing functional, physical and emotional scales
Voice quality of life | Post-operative 2 weeks
  Voice Handicap Index - 30 assessing functional, physical and emotional scales
Voice quality of life | Post-operative 6 months
  Voice Handicap Index - 30 assessing functional, physical and emotional scales
Swallowing quality of life | Post-operative day 1
  MD Anderson dysphagia inventory (MDADI)
Swallowing quality of life | Post-operative 2 weeks
  MD Anderson dysphagia inventory (MDADI)
Swallowing quality of life | Post-operative 6 months
  MD Anderson dysphagia inventory (MDADI)
Complication rate and types | Post-operative 2 weeks
  Lower lip numbness, skin bruising or injury, wound infection, vocal cord paralysis, temporary hypoparathyroidism
Complication rate and types | Post-operative 6 months
  Lower lip numbness, vocal cord paralysis, permanent hypoparathyroidism

SECONDARY OUTCOMES:
Inpatient stay | An average of 0-2 days after the operation
  Number of days of inpatient stay
Operative time | Intra-operatively
  Minutes
Blood loss | Intra-operatively
  Volume
Rate of conversion to open surgery | Intra-operatively
  Percentage of conversion

CONTACTS AND LOCATIONS:
Overall Officials: Jason YK Chan, Study Director — Department of Otorhinolaryngology, Head and Neck Surgery, The Chinese University of Hong Kong; Zenon Yeung, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery, The Chinese University of Hong Kong
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, United Christian Hospital and Tseung Kwan O Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No